CLINICAL TRIAL: NCT00002498
Title: CMF AND MITOXANTRONE IN ELDERLY PATIENTS WITH ADVANCED BREAST CANCER, A RANDOMIZED PHASE II STUDY
Brief Title: Combination Chemotherapy Compared With Mitoxantrone in Treating Older Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077804; DUT-KWF-CKVO-9008; EU-92006
Record Dates: First submitted 1999-11-01; First posted 2004-08-23 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2000-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Fluorouracil; Methotrexate; Mitoxantrone

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: fluorouracil
Drug: methotrexate
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs in different combinations may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of cyclophosphamide, methotrexate, and fluorouracil with mitoxantrone in treating older patients with recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and duration of response of elderly patients with advanced breast cancer treated with first-line chemotherapy with mitigated "classical" CMF (cyclophosphamide/methotrexate/fluorouracil) vs. mitoxantrone (DHAD). II. Define the morbidity of CMF and DHAD in elderly patients. III. Determine quality of life in these patients.

OUTLINE: This is a randomized study. Patients are stratified by participating institution. The first group receives oral cyclophosphamide on days 1 through 14 and intravenous methotrexate and fluorouracil on days 1 and 8. Courses repeat every 4 weeks for a maximum of 6 courses. The second group receives intravenous mitoxantrone every 3 weeks for a maximum of 8 courses. Concomitant therapy with hepatotoxic or nephrotoxic drugs (e.g., NSAIDs) or corticosteroids (even as antiemetics) is not permitted in either group. Radiotherapy is allowed provided no more than 50% of the bone marrow is irradiated and at least 1 indicator lesion is unirradiated. Patients who complete therapy are followed every 3 months until disease progression.

PROJECTED ACCRUAL: 60 patients will be accrued over approximately 1 year. If extreme differences between arms exist after entry of 30 patients, accrual may be stopped early.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, progressive, recurrent or metastatic breast cancer in patients over 70 years of age Measurable or evaluable disease required, including: Lesions of the mediastinum, retroperitoneum, or liver at least 3 cm in diameter on CT scan or ultrasound The following are not considered measurable or evaluable: Lymphedema Hilar enlargement Pleural effusion Ascites Bone marrow infiltration Osteoblastic skeletal lesion No CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Over 70 Sex: Not specified Menopausal status: Postmenopausal Performance status: WHO 0-2 Hematopoietic: WBC at least 3,000 Platelets at least 100,000 Hepatic: Bilirubin less than 1.4 mg/dL (25 micromoles/L) Renal: Creatinine clearance (calculated) greater than 50 mL/min in patients weighing at least 45 kg and measured creatinine clearance at least 50 mL/min in patients weighing less than 45 kg Cardiovascular: No congestive heart failure No myocardial infarction within 6 months No severe arrhythmia No complete bundle branch block Other: No active uncontrolled infection No mental disorders that may preclude patient follow-up No second malignancy except: Adequately treated basal cell carcinoma of the skin Adequately treated in situ carcinoma of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for advanced disease At least 1 year since prior adjuvant chemotherapy Endocrine therapy: At least 4 weeks since prior estrogens, androgens, and progestins Tamoxifen or aminoglutethimide allowed with no waiting period if disease progresses Recovery from prior hormonal therapy for metastatic disease required Radiotherapy: Prior radiotherapy allowed provided: Evaluable disease exists outside of treatment field No greater than 50% of bone marrow was irradiated Surgery: Not specified

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 1992-07

CONTACTS AND LOCATIONS:
Overall Officials: Marianne A. Nooij, MD, Study Chair — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - St. Radboud University Hospital, Nijmegen